CLINICAL TRIAL: NCT01535547
Title: Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Tacrolimus: A Phase 1, Open Label, Sequential Study in Healthy Adult Subjects
Brief Title: Drug Interaction Study of Isavuconazole and Tacrolimus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0021
Record Dates: First submitted 2012-02-15; First posted 2012-02-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of Tacrolimus; Healthy Volunteers
Keywords: isavuconazole; tacrolimus; Healthy Volunteers; BAL8557
MeSH Terms: interventions — isavuconazole; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- isavuconazole and tacrolimus (Experimental)
  Interventions: Drug: isavuconazole; Drug: tacrolimus

INTERVENTIONS:
Drug: isavuconazole — oral
  Other Names: BAL8557; BAL4815
Drug: tacrolimus — oral
  Other Names: Prograf; FK506

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics (PK) of tacrolimus after single dose administration.

DETAILED DESCRIPTION:
Subjects will receive a single dose of tacrolimus on Day 1 followed by a 15 day wash-out period (time from tacrolimus dosing to isavuconazole dosing).

On Days 16 and 17, isavuconazole will be dosed three times daily (TID). TID doses will be administered 8 hours apart. On Days 18 through 28 isavuconazole will be administered once daily (QD). All subjects will be administered a single dose of tacrolimus on Day 20. A follow up visit will occur approximately 7 days after the last dose of isavuconazole. Blood samples for pharmacokinetics will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject must weigh at least 45 kg and have a body mass index (BMI) of 18 to 32 kg/m2, inclusive
* The subject has a normal 12-lead electrocardiogram (ECG)
* The subject's clinical laboratory test results are within normal limits
* Results for aspartate aminotransferase (AST), alanine aminotransferase (ALT) and total bilirubin must be within the normal range
* If female, the subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years without menses), or using a medically acceptable double barrier method to prevent pregnancy and agrees to continue using this method from Screening until three weeks after the follow up visit at the end of study; and is not lactating or pregnant as documented by negative serum pregnancy tests
* If male, the subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy during the study period and for three weeks after the follow up visit at the end of the study

Exclusion Criteria:

* Any clinically significant disease history of the following systems: pulmonary, gastrointestinal, cardio-vascular (including a history of clinically significant arrhythmia or clinically significant conduction delays on ECG), hepatic, neurological, psychiatric, renal, genitourinary, endocrine, metabolic, dermatologic, immunologic, hematologic, or malignancy excluding non melanoma skin cancer
* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* History of tuberculosis or exposure to anyone known or suspected to have tuberculosis or any illness that might confound the results of the study or pose additional risk in administering study drug to the subject
* The subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic admission
* The subject has received a vaccination within the last 30 days prior to study drug administration or plans to receive any vaccinations within 2 weeks after the last dose of study drug
* The subject has a positive result for hepatitis B surface antigen, hepatitis C antibodies, or QuantiFERON®-TB Gold test(s) or is known to be positive for human immunodeficiency virus
* The subject has a known or suspected allergy to any of the components of the trial products including tacrolimus or the azole class of compounds or a history of multiple and/or severe allergies to drugs or foods or a history of hypersensitivity to polyoxyl 60 hydrogenated castor oil, or a history of severe anaphylactic reactions
* The subject is a smoker (any use of tobacco or nicotine containing products) in the last 6 months
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to study drug administration, or over-the-counter medication within 1 week prior to Day -1, with the exception of acetaminophen up to 2 g/day
* The subject has received an experimental agent within 30 days or 5 half-lives, whichever is longer, prior to Day -1
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission
* The subject has taken part in strenuous exercise within 3 days before dosing in this trial
* The subject anticipates an inability to abstain from caffeine or alcohol use for 48 hours prior to clinic admission and throughout the duration of the study; or from grapefruit, grapefruit juice, star fruit, or Seville oranges or any products containing these items from 72 hours prior to clinic admission and throughout the duration of the study
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, or a positive drug screen
* The subject has any other condition which precludes the subject's participation in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetic (PK) variables for tacrolimus (in whole blood) : AUClast , AUCinf, Cmax, tmax , Vz /F, CL/F and t1/2 | Days 1 and 20
  Area under the curve (AUC) from time of dosing to last quantifiable concentration (AUClast ), AUC from time 0 extrapolated to infinity (AUCinf), and maximum concentration (Cmax), time to attain Cmax (tmax) , apparent volume of distribution (Vz /F), apparent body clearance after oral dosing (CL/F) and apparent terminal elimination half-life (t1/2 ).
PK variable for isavuconazole (in plasma): trough concentration (Ctrough) | Days 18 and Days 22 through 29
Composite of PK variable for isavuconazole (in plasma): trough concentration (Ctrough), AUC during the time interval between consecutive dosing (AUCtau), maximum concentration (Cmax),and time to attain Cmax (tmax) | Days 19 and 20

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Covance, Madison, Wisconsin, United States